CLINICAL TRIAL: NCT02782052
Title: Bronchodilator's Effects on Exertional Dyspnoea in Pulmonary Arterial Hypertension
Acronym: BD-HTAP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P130906; 2014-002590-10 (EudraCT Number)
Record Dates: First submitted 2016-05-17; First posted 2016-05-25 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; spirometry; dynamic lung hyperinflation; bronchodilator; dyspnoea; Idiopathic; heritable; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Dyspnea | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nebulized ipratropium bromide (Experimental): Administration in a random order nebulized ipratropium bromide at V3 or V4 or V5
  Interventions: Drug: Nebulized ipratropium bromide
- Nebulized combination ipratropium bromide with salbutamol (Experimental): Administration in a random order combination Ipratropium bromide and Salbutamol at V3 or V4 or V5
  Interventions: Drug: Nebulized combination ipratropium bromide with salbutamol
- Placebo (Placebo Comparator): Administration in a random order placebo at V3 or V4 or V5
  Interventions: Drug: Nebulized Placebo

INTERVENTIONS:
Drug: Nebulized ipratropium bromide — Administration at V3 or V4 or V5 in a random order:
  * Placebo (P; sterile 0.9% sodium chloride solution)
  * Or nebulized ipratropium bromide (IB; 0.5mg/2mL) alone
  * Or nebulized combination ipratropium bromide with salbutamol (IB+SALB; 0.5mg/2mL + 2.5mg/2.5mL).
  Arms: Nebulized ipratropium bromide
Drug: Nebulized combination ipratropium bromide with salbutamol — Administration at V3 or V4 or V5 in a random order:
  * Placebo (P; sterile 0.9% sodium chloride solution)
  * Or nebulized ipratropium bromide (IB; 0.5mg/2mL) alone
  * Or nebulized combination ipratropium bromide with salbutamol (IB+SALB; 0.5mg/2mL + 2.5mg/2.5mL).
  Arms: Nebulized combination ipratropium bromide with salbutamol
Drug: Nebulized Placebo — Administration at V3 or V4 or V5 in a random order:
  * Placebo (P; sterile 0.9% sodium chloride solution)
  * Or nebulized ipratropium bromide (IB; 0.5mg/2mL) alone
  * Or nebulized combination ipratropium bromide with salbutamol (IB+SALB; 0.5mg/2mL + 2.5mg/2.5mL).
  Arms: Placebo

SUMMARY:
Activity-related dyspnoea appears to be the earliest and the most frequent complaint for which patients with PAH seek medical attention. This symptom progresses relentlessly with time leading invariably to avoidance of activity with consequent skeletal muscle deconditioning and an impoverished quality of life. Unfortunately, effective management of this disabling symptom awaits a better understanding of its underlying physiology. Our team has recently showed that PAH patients may exhibit reduced expiratory flows at low lung volumes at spirometry (namely instantaneous forced expiratory flows measured after 50% and 75% of the FVC has been exhaled [FEF50% and FEF75%] lower than predicted), despite a preserved forced expiratory volume in 1 second/forced vital capacity ratio (FEV1/FVC) . Several studies have shown that such a finding ("small airway disease") could be common in certain PAH cohorts, have either related it to incidental descriptions of airway wall thickening with lymphocytic infiltration in PAH or proposed several other speculative explanatory mechanisms, either biological or mechanical. Whatever its cause, reduced expiratory flows at low lung volumes imply that the operating tidal volume (VT) range becomes closer than normally to residual volume (RV) mostly through an increase in RV (elevated residual volume/total lung capacity ratio, RV/TLC). The reduced difference between forced and tidal expiratory flows promotes dynamic lung hyperinflation [i.e., a progressive increase in end-expiratory lung volume (EELV)] under conditions of increased ventilatory demand. Dynamic lung hyperinflation (DH) is well known to have serious sensory consequences, i.e., increase in dyspnoea intensity, as clearly shown in patients with chronic obstructive pulmonary disease and chronic heart failure. The aim of this study is to evaluate whether administration of inhaled BDs (β2-agonist and/or anticholinergic), as add-ons to vasodilators, would be beneficial to PAH patients by reducing and/or delaying the rate of onset of DH, thus ameliorating the exertional symptoms in patients with stable PAH undergoing high-intensity constant work-rate (CWR) cycle endurance test.

This is a randomised double-blind placebo-controlled crossover study. Design: 5 visits; V1: screening, familiarization, incremental cardiopulmonary exercise testing (CPET); V2: constant work-rate (CWR-CPET); V3, V4 and V5: CWR-CPET after intervention, in a random order: Placebo (P), Ipratropium Bromide (IB), Ipratropium Bromide + Salbutamol (IB+SALB).

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH), defined as a mean pulmonary arterial pressure (mPAP) of ≥25 mmHg at rest and pulmonary arterial wedge pressure ≤15 mmHg, is consistently associated with reduced exercise capacity and intolerable dyspnoea (respiratory difficulty) on exertion. Dyspnoea is a complex multifaceted and highly personalized sensory experience, the source and mechanisms of which are incompletely understood. Activity-related dyspnoea appears to be the earliest and the most frequent complaint for which patients with PAH seek medical attention. This symptom progresses relentlessly with time leading invariably to avoidance of activity with consequent skeletal muscle deconditioning and an impoverished quality of life. Unfortunately, effective management of this disabling symptom awaits a better understanding of its underlying physiology. Previous studies on mechanisms of exertional dyspnoea in PAH have largely and mostly focused on the cardiovascular determinants of respiratory discomfort. However, respiratory mechanics abnormalities could contribute to exertional dyspnoea in these patients. For instance, PAH patients may exhibit reduced expiratory flows at low lung volumes at spirometry (namely instantaneous forced expiratory flows measured after 50% and 75% of the FVC has been exhaled [FEF50% and FEF75%] lower than predicted), despite a preserved forced expiratory volume in 1 second/forced vital capacity ratio (FEV1/FVC). Several studies have shown that such a finding ("small airway disease") could be common in certain PAH cohorts, have either related it to incidental descriptions of airway wall thickening with lymphocytic infiltration in PAH or proposed several other speculative explanatory mechanisms, either biological or mechanical. Whatever its cause, reduced expiratory flows at low lung volumes imply that the operating tidal volume (VT) range becomes closer than normally to residual volume (RV) mostly through an increase in RV (elevated residual volume/total lung capacity ratio, RV/TLC). The reduced difference between forced and tidal expiratory flows promotes dynamic lung hyperinflation [i.e., a progressive increase in end-expiratory lung volume (EELV)] under conditions of increased ventilatory demand. Dynamic lung hyperinflation (DH) increases the mechanical inspiratory load that the respiratory muscles must overcome to produce ventilation (V'E), places the diaphragm at mechanical disadvantage, and reduces the ability of VT to expand appropriately during exercise, thus imposing "restrictive" mechanics: VT is therefore truncated from below by the increasing EELV and constrained from above by the total lung capacity (TLC) envelope and the relatively reduced inspiratory reserve volume (IRV). Dynamic hyperinflation-induced critical mechanical constraint of VT expansion has serious sensory consequences, i.e., increase in dyspnoea intensity, as clearly shown in patients with chronic obstructive pulmonary disease and chronic heart failure.

In this regard, our team has recently confirmed that small airway dysfunction at spirometry exists in the majority of PAH patients (60%) despite preserved FEV1/VC, and that this promotes the development of DH under the increased ventilatory demand in response to physical task: in fact, during the accelerated ventilatory response to exercise, 60% of PAH patients did increase their EELV (i.e., DH) by an average of 0.50L from rest to peak exercise, whereas age- and sex-matched healthy subjects did decrease it by an average of 0.45L. Similar levels of DH have been reported in healthy subjects between 40 and 80 years of age, patients with mild-to-severe COPD, CHF, and recently also in a heterogeneous group of patients with precapillary pulmonary hypertension, but at much lower V'E and work-rate than in our more homogeneous group of PAH patients. Our team did also show that DH had serious sensory consequences for PAH patients. DH imposed severe mechanical constraints on VT expansion during exercise on a background of progressively increasing central neural drive: VT was truncated from below by the increasing EELV and constrained from above by the TLC envelope and the relatively reduced IRV. It is generally accepted that in this setting dyspnoea results from the conscious awareness of the increasing disparity between respiratory effort (or neural drive to breathe) and simultaneous thoracic volume displacement. The notion that DH and the subsequent constraint of VT expansion contributed to exertional dyspnoea was bolstered by the strong inverse correlation between dyspnoea intensity and both the increase dynamic EELV/TLC(%) (R=0.70, p<0.05) and the reduced IRV/TLC(%) (R=-0.78, p<0.05) at a standardized exercise stimulus.

Our team was able, for the first time, to clearly demonstrate that an abnormal mechanics of breathing (dynamic lung hyperinflation and the attendant constraint of VT expansion) played an important role in dyspnoea causation in PAH during cycle exercise. When increased ventilation/perfusion mismatching is superimposed on pre-existing abnormal airway function, greater troublesome exertional symptoms are the result. This finding opens up new horizons for research in the field of dyspnoea mechanisms in PAH: if investigator treats and ameliorates the "lung function" (i.e., the respiratory mechanics abnormalities"), then our team could be able to improve the troublesome exertional symptoms that curtail daily-living activities of PAH patients. The corollary of this is that any therapeutic intervention that effectively reduces and/or delays the rate of onset of DH-induced critical ventilatory constraints, such as administration of inhaled bronchodilators (BDs) as add-ons to vasodilators, should have a positive effect on symptom perception in selected patients with stable PAH. Determining the magnitude of this effect will be the object of the planned experiments. However, it should be borne in mind that the relationship between dyspnoea intensity and the severity of respiratory abnormalities is not linear, but rather exponential. In other words, when a given disease is already responsible for a very intense dyspnoea, a small additional deterioration directly or indirectly related to the disease can make dyspnoea intolerable. Therefore, even small BDs-induced changes in respiratory mechanics could have major effects on dyspnoea intensity on exertion in selected PAH patients, which would undoubtedly have a major impact on their quality of life and their ability to perform daily-living activities.

Hypothesis for the research What is the potential mechanism by which BDs would be able to ameliorate the exertional symptoms in patients with stable PAH, and, which BDs would be the best candidate in achieving that? Regardless of the BDs administered, our team anticipates that the potential mechanism by which BDs are able to ameliorate the exertional symptoms in patients with stable PAH would be the reduction and/or delay of the rate of onset of DH-induced critical ventilatory constraints during exercise. In contrast, the nature of the specific BD (β2-agonist or anticholinergic) would be important in determining the mechanism by which the reduction in DH-induced critical ventilatory constraints can be achieved. BDs have been extensively studied in COPD patients, and to less extent in CHF patients. Little is known in PAH patients. Spiekerkoetter and colleagues have recently pointed out that inhaled β2-agonists are able to cause a mild but significant increase in resting FEV1, FEF50% and FEF75% in PAH patients. They also showed that inhalation of β2-agonists determined a significant increase in resting cardiac output accompanied by an increase in stroke volume and a decrease in pulmonary and systemic vascular resistance, in the presence of no change in heart rate. To date, no information is available on the effects of inhaled β2-agonists on the ventilatory, mechanical and perceptual responses to exercise in PAH patients. It can be argued that β2-agonists may reduce and/or delay the rate of onset of DH-induced critical ventilatory constraints by 1) reducing the ventilatory demand in response to exercise, and/or by 2) modifying the shape and limits of the maximal flow-volume loop (MFVL). In the first case, the improved cardiac function and concurrent ventilation-perfusion relations following β2-agonists would reduce the ventilatory demand, thereby reducing the rate of DH and enhancing VT expansion during exercise. This, in turn, would be expected to reduce the perceived exertional dyspnoea, as clearly shown in patients with COPD following BDs. In the second case, β2-agonists would increase the maximal volume-corrected expiratory flow rates in the effort-independent mid-volume range where tidal breathing occurs (i.e., increase in FEF50% and FEF75%), as it has been shown in CHF. This means that PAH patients would now accomplish the required alveolar ventilation at a lower operating lung volume and, therefore, at a reduced oxygen cost of breathing during exercise. The corollary of this will be that PAH patients would increase their end-expiratory lung volume (i.e., DH) to less extent after inhalation of β2-agonist than before, and this is likely to have salutary sensory consequences (i.e., reduction in dyspnoea intensity) for patients with PAH, as clearly shown in patients with COPD. Inhaled anticholinergic agents have not yet been studied, neither at rest nor during exercise in PAH. Inhalation of anticholinergic agents would increase the maximal volume-corrected expiratory flow rates in the effort-independent mid-volume range where tidal breathing occurs, without interfering with the cardiac and pulmonary vascular functions, as it has been shown in patients with CHF. The attendant increase in FEF50% and FEF75% (where tidal breathing occurs) following inhaled anticholinergic agents would cause VT to be accommodated at a lower operating lung volume, thus reducing the extent of DH and the concurrent ventilatory constraints imposed by the accelerated ventilatory response to exercise. This, in turn, is likely to have salutary sensory consequences (i.e., reduction in dyspnoea intensity) for patients with PAH. The interest of our study in dyspnoea evaluation after BDs in PAH patients is, therefore, evident and appealing, for at least two reasons: 1) there is no information in the literature about the effect of pharmacological interventions on dyspnoea intensity (measured by Borg score) during cycle exercise in PAH population, and 2) investigators do not know how much will the dyspnoea intensity (measured by Borg score) change after BD administration in PAH population because no Minimally Clinically Important Difference (MCID) has been established for measurements of dyspnoea intensity. Nonetheless, based on COPD studies, short-term post-intervention changes in dyspnoea intensity of ~1 Borg unit at a standardized exercise time or V'E appear to be clinically meaningful, therefore our team can assume that this MCID may also apply to PAH patients undergoing cycle exercise testing after BD interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (> 18 years old);
2. With signed informed consent;
3. Affiliated to social security system;
4. With idiopathic or heritable PAH , diagnosed according to the current evidence-based clinical practice guidelines;
5. Irrespective of the treatment received;
6. Clinically stable during the 3 preceding months and the entire duration of the project;
7. With CPET scheduled within the frame of their clinical follow-up at the reference center.

Exclusion Criteria:

1. Pregnant women;
2. Past or current tobacco-smoking history;
3. A spirometric evidence of an obstructive ventilatory defect as defined by a reduced FEV1/VC ratio below the 5th percentile of the predicted value;
4. A FEF75% >60% of predicted normal values at spirometry;
5. A TLC below the 5th percentile of the predicted value;
6. A body mass index >30 kg.m-2;
7. Use of supplemental oxygen;
8. PAH induced by drugs and toxins;
9. PAH associated with other conditions, including connective tissue diseases, congenital heart diseases, portal hypertension, and HIV infection;
10. Chronic thromboembolic pulmonary hypertension;
11. Other respiratory, cardiac and other diseases that could contribute to dyspnoea or exercise limitation;
12. Contraindications to clinical exercise testing, such as NYHA functional class IV, syncope and others;
13. Specific contraindications (precautions and drug interactions) to the administration of IB or IB+SALB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-10 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of 1.0 unit of dyspnoea intensity (on a Borg scale) between pre-dose and post-dose BD measured at a standardized time (iso-time) or V'E (iso-V'E) | At two month (V3), three month (V4) and three months (V5)
  At the end of CWR-CPET, the sensory-perceptual and affective dimensions of dyspnoea will be evaluated with Multidimensional Dyspnoea Profile (MDP) questionnaire.

SECONDARY OUTCOMES:
Difference (BDs versus placebo) in CWR endurance time (60 seconds difference) will be also evaluated as potential index of improved exercise tolerance | At two month (V3), three month (V4) and three months (V5)
  Change (increase) of at least 60 seconds in CWR-CPET endurance time between pre-dose and post-dose BD measured at the end of CWR bouts.

IPD SHARING:
Plan to Share IPD: No